CLINICAL TRIAL: NCT00920283
Title: Randomized Comparison Between Two Cobalt-Chromium Balloon Expandable Stents for the Treatment of De Novo Coronary Artery Lesions
Brief Title: COMPETE: A Clinical Evaluation of Chrono Carbostent Carbofilm™ Coated Stent
Acronym: COMPETE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: CID - Carbostent & Implantable Devices (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: C10901
Record Dates: First submitted 2009-06-12; First posted 2009-06-15 (Estimated); Last update posted 2018-05-07 (Actual); Status verified 2018-05

CONDITIONS: Coronary Atherosclerotic Disease; Coronary Occlusive Diseases; Coronary Artery Diseases; Myocardial Ischemia; Coronary Stenosis
Keywords: Stents; Bare Metal Stents; PCI; Coronary Artery Disease; Coronary Artery Stenosis; Stent Thrombosis; Vascular Disease; Myocardial Ischemia
MeSH Terms: conditions — Coronary Artery Disease; Myocardial Ischemia; Coronary Stenosis; Vascular Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Chrono Carbostent Carbofilm™ Coated Coronary Stent (Experimental)
  Interventions: Device: Chrono Carbostent Carbofilm™ Coated Coronary Stent
- Driver, Cobalt Alloy Coronary Stent (Active Comparator)
  Interventions: Device: Driver Cobalt Alloy Coronary Stent

INTERVENTIONS:
Device: Chrono Carbostent Carbofilm™ Coated Coronary Stent
  Arms: Chrono Carbostent Carbofilm™ Coated Coronary Stent
Device: Driver Cobalt Alloy Coronary Stent
  Arms: Driver, Cobalt Alloy Coronary Stent

SUMMARY:
The COMPETE study is a prospective,randomized,two-arm multi-center clinical trial comparing two commercially available coronary stents: Chrono Carbostent Carbofilm™ Coated vs Driver/Micro-Driver Coronary Stent System. In this study, 204 subjects will be included (2:1 randomization Chrono:Driver/Micro Driver) in 6 Italian sites.

ELIGIBILITY:
Inclusion Criteria:

* Patients with clinical evidence of ischemic heart disease;
* No clinical and ECG changes suggestive of ongoing acute infarction;
* De novo lesion > 50% and <100% diameter stenosis (DS) in native coronary vessels TIMI flow of >= 1.
* Reference diameter > 2.5 mm or < 4.0 mm;
* Patients with a maximum of two coronary lesions to be treated with a maximum of 2 study stents;

Exclusion Criteria:

* Lesion length > 30 mm;
* Significant (>50%) stenosis proximal or distal to the target lesions that might impede run off;
* Lesions located in saphenous vein graft;
* Lesions located in unprotected left main;
* Presence of > 40% stenosis in the left main;
* Ostial lesion;
* Lesion located in a bifurcation;
* Target lesion with visible thrombus;
* Chronic total occlusion;
* Treatment of restenotic lesions;
* Previous implantation of a stent (BMS/DES) in the target vessel.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 205 (Actual)
Dates: Start 2009-07 (Actual); Primary Completion 2012-12 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
in-stent late lumen loss (LLL) | 180 days

SECONDARY OUTCOMES:
Angiographic binary restenosis (diameter stenosis ≥50%) | 180 days
Clinical Composite Endpoints: - Cardiac death/ MI - Cardiac death / Target vessel MI / (Clinically indicated) TLR* - All death / MI / all repeat revascularization** *Device oriented composite endpoint **Patient oriented composite endpoint | 30 days, 180 days, 1 year
Stent Thrombosis | acute, 30 days, 180 days, 1 year
Acute success (Device and Procedural success) | acute

CONTACTS AND LOCATIONS:
Overall Officials: Flavio Airoldi, Dr, Principal Investigator — Multimedica IRCCS, Sesto SG (MI) Italy
Locations (6):
- Italy (6):
  - Maria Cecilia Hospital, Cotignola, Ravenna
  - Cardinal Massaia Hospital, Asti
  - Azienda Ospedaliera Policlinico di Modena, Modena
  - Ospedale Civile S.Agostino-Estense-Baggiovara, Modena
  - Azienda Ospedaliera Universitaria, Roma
  - Ospedale Civile Maggiore- Borgo Trento, Verona